CLINICAL TRIAL: NCT00522392
Title: Randomized Phase III Trial of Consolidation Therapy With Bortezomib (Velcade®)-Lenalidomide (Revlimid®) -Dexamethasone (VRD) Versus Bortezomib (Velcade®)-Dexamethasone (VD) for Patients With Multiple Myeloma Who Have Completed a Dexamethasone Based Induction Regimen
Brief Title: Bortezomib and Dexamethasone With or Without Lenalidomide in Treating Patients With Multiple Myeloma Previously Treated With Dexamethasone
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00521; NCI-2009-00521 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E1A05 (Other: Eastern Cooperative Oncology Group (ECOG)); U10CA021115 (NIH); U10CA180820 (NIH)
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Results first posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-05

CONDITIONS: Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
Keywords: Consolidation therapy; First-line therapy; Proteasome inhibitor; Thalidomide analogue; Quality of life
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (VRD) (Experimental): Patients were given consolidation therapy for 8 cycles (1 cycle = 21 days) with the combination bortezomib, dexamethasone and lenalidomide. Patients received each cycle: the standard dose of bortezomib (1.3 mg/m2) on days 1, 4, 8 and 11; fixed dose of lenalidomide at 15 mg orally on days 1-14; and 3 days of dexamethasone at 40 mg total dose per day given on days 1, 8 and 15. Aspirin 325 mg/day orally on days 1-21 of each cycle was required unless the patient was treated with alternate prophylaxis of either low molecular weight heparin or coumadin.
  Interventions: Drug: bortezomib; Drug: lenalidomide; Drug: dexamethasone
- Arm B (VD) (Active Comparator): Patients were given consolidation therapy for 8 cycles (1 cycle = 21 days) with the combination bortezomib plus dexamethasone. Patients received each cycle: the standard dose of bortezomib (1.3 mg/m2) on days 1, 4, 8 and 11 and 3 days of dexamethasone at 40 mg total dose per day given on days 1, 8 and 15.
  Interventions: Drug: bortezomib; Drug: dexamethasone

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: PS-341; LDP-341; MLN-341; VELCADE
Drug: lenalidomide — Given PO
  Other Names: CC-5013; CDC-501; Revlimid® (formerly Revimid®)
  Arms: Arm A (VRD)
Drug: dexamethasone — Given PO
  Other Names: Decadron; Hexadrol; Dexameth; Dexone; DXM

SUMMARY:
This randomized phase III trial compares bortezomib, dexamethasone, and lenalidomide with bortezomib and dexamethasone to see how well they work in treating patients with multiple myeloma previously treated with dexamethasone. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Lenalidomide may stimulate the immune system in different ways and stop cancer cells from growing. It is not yet known whether giving bortezomib and dexamethasone is more effective with or without lenalidomide in treating multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression-free survival (PFS) for two consolidation regimens: bortezomib, lenalidomide, and dexamethasone (VRD) versus bortezomib and dexamethasone (VD) only.

SECONDARY OBJECTIVES:

I. To determine the incremental ability of VRD versus VD in attaining a complete response or a very good partial response (VGPR) in patients receiving induction therapy with a dexamethasone based induction regimen.

II. To compare the overall survival, measured from the time of study entry.

III. Evaluate response rate and PFS according to cytogenetic category (by gene expression and fluorescence in situ hybridization [FISH]).

IV. To evaluate the toxicity of the two regimens.

V. To compare quality of life (QOL) based on the Functional Assessment of Cancer Therapy (FACT)-Neurotoxicity (Ntx) Trial Outcome Index (TOI) of patients receiving VD to those receiving VRD from registration to 6 months post consolidation treatment.

VI. To examine the impact of differential treatment response (PFS), if observed, on QOL based on the FACT-Ntx TOI up to 12 months post consolidation treatment.

VII. To obtain prospective data on multiple myeloma specific QOL attributes.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive bortezomib at 1.3 mg/m2 intravenously (IV) on days 1, 4, 8, and 11, lenalidomide orally (PO) once daily (QD) at 15 mg on days 1-14, and dexamethasone at 40 mg total dose per day PO QD on days 1, 8, and 15. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive bortezomib at 1.3 mg/m2 IV on days 1, 4, 8, and 11 and dexamethasone at 40 mg total dose per day PO QD on days 1, 8, and 15. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then every 12 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic multiple myeloma, that was symptomatic at time of initial diagnosis, but may be asymptomatic at the time of registration based on induction therapy
* For the original diagnosis of myeloma, patients must have met the following criteria at one point in their disease course: bone marrow plasmacytosis (>10% plasma cells or sheets of plasma cells) or a biopsy proven plasmacytoma, and evidence of end-organ damage due to multiple myeloma including anemia, hypercalcemia, bone disease (lytic bone lesions or pathologic fractures) or renal dysfunction.
* Patients may have prior exposure to bortezomib
* Patients must have received a minimum of 1 cycle, maximum of 6 cycles, of a dexamethasone-based regimen; patient must not have experienced progressive disease on such therapy
* The following induction regimens were considered adequate for enrollment: dexamethasone alone; vincristine, doxorubicin and dexamethasone; thalidomide and dexamethasone; lenalidomide and dexamethasone; liposomal doxorubicin and dexamethasone; the combination of any of the above agents and dexamethasone; or cyclophosphamide, lenalidomide and dexamethasone
* Patients must have received the minimum cumulative dose of dexamethasone of 160 mg (sum of induction treatment) with no maximum dose specified
* Patients must have been offered and refused front-line stem cell transplant OR not have been eligible for front-line stem cell transplant.
* Bone marrow aspiration and/or biopsy must be obtained =< 28 days prior to randomization
* All tests below must be performed =< 28 days prior to randomization:

  * Kappa free light chain mg/dL
  * Lambda free light chain mg/dL
  * Serum M-protein by serum protein electrophoresis (SPEP)
  * Urine M-protein light chain excretion by urine protein electrophoresis (UPEP)
* Adequate laboratory levels within 7 days prior to randomization: hemoglobin > 7 g/dL, platelet count > 75,000 cells/mm^3, absolute neutrophil count > 1000 cells/mm^3, creatinine < 2.5 mg/dL, creatinine clearance (measured or calculated) >= 60 mL/min, direct bilirubin =< 1.5 mg/dL, serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) and serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2.5 times the upper limit of normal
* Patients may be receiving bisphosphonates or erythropoietin growth factors (erythropoietic agents) for multiple myeloma
* Prior palliative and/or localized radiation therapy is permitted, provided at least 14 days have passed from date of last radiation therapy to date of randomization
* Patients must be willing and able to take prophylaxis with either aspirin at 325 mg/day or alternative prophylaxis with either low molecular weight heparin or coumadin (patients with prior deep vein thrombosis [DVT] are eligible provided they remain on the anticoagulation regimen that was prescribed for treatment of the DVT throughout the protocol therapy)
* Patients must be competent to understand the study as explained in the consent form
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Sexually active males must be willing to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking lenalidomide, and for 4 weeks after stopping treatment
* Patients with a history of prior malignancy are eligible provided there is no active malignancy and a low expectation of recurrence within 6 months
* Age >=18 years

Exclusion Criteria:

* More than 8 weeks from the last day of last cycle of induction treatment
* Active, uncontrolled seizure disorder; seizures in the last 6 months
* Uncontrolled inter-current illness that would limit compliance with the study including uncontrolled hypertension, symptomatic congestive heart failure, unstable angina, uncontrolled cardiac arrhythmia, uncontrolled psychiatric illness or social situation, prior history of Stevens Johnson syndrome
* Grade 2 or higher peripheral neuropathy by Common Terminology Criteria for Adverse Events (CTCAE) version 3.0
* Active, uncontrolled infection
* Smoldering myeloma or monoclonal gammopathy of undetermined significance
* Pregnant or nursing women were not eligible. Women of child-bearing potential unwilling to use a dual method of contraception and men who were unwilling to use a condom were not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-09; Primary Completion 2012-08 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Fonseca, M.D., Study Chair — Mayo Clinic
Locations (276):
- United States (275):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Northbay Cancer Center, Fairfield, California
  - Kaiser Permanente, San Diego, California
  - Stanford University Hospitals and Clinics, Stanford, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Mayo Clinic in Florida, Jacksonville, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Saint Anthony's Health, Alton, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Alexian Brothers Medical and Cancer Center, Elk Grove Village, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Medical Center, Waterloo, Iowa
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Union Hospital of Cecil County, Elkton MD, Maryland
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Duluth Clinic CCOP, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Capital Regional Medical Center, Jefferson City, Missouri
  - Ozark Health Ventures LLC dba Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Good Samaritan Hospital, Kearney, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Kings County Hospital, Brooklyn, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - University Hospital of Brooklyn, Brooklyn, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Adirondack Cancer Center, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - Montefiore Medical Center, The Bronx, New York
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Adventist Medical Center, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Mainline Health CCOP, Wynnewood, Pennsylvania
  - McLeod Regional Medical Center, Florence, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Columbia Basin Hematology and Oncology PLLC, Kennewick, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - The Schiffler Cancer Center of Wheeling Hospital, Wheeling, West Virginia
  - Wheeling Hospital, Wheeling, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- University Of Pretoria, Pretoria, South Africa

REFERENCES:
- [Background] Fonseca R, Rajkumar SV. Consolidation therapy with bortezomib/lenalidomide/ dexamethasone versus bortezomib/dexamethasone after a dexamethasone-based induction regimen in patients with multiple myeloma: a randomized phase III trial. Clin Lymphoma Myeloma. 2008 Oct;8(5):315-7. doi: 10.3816/CLM.2008.n.046. PMID 18854289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG member institutions between September 6, 2007 and May 7, 2010.
Period: Overall Study
Arm/Group | Arm A (VRD) | Arm B (VD)
Started | 23 | 25
Pts w/ Measurable Disease at Baseline | 16 | 16
Pts w/ QOL Assessments Complete | 12 | 8
Completed | 15 | 12
Not Completed | 8 | 13
Not completed — Disease progression | 0 | 3
Not completed — Adverse Event | 7 | 7
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (VRD) | Arm B (VD) | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Continuous [Median (Full Range); unit: years] | 64 [33 to 76] | 65 [33 to 74] | 65 [33 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 15 | 12 | 27
Region of Enrollment [Number; unit: participants]
  United States | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was defined as the time from randomization to the earliest documentation of disease progression (PD) or death. If a patient died without evidence of PD, the patient was considered an event if death occurred within 3 months of the last disease assessment. Patients who died outside of the specified interval or patients who were alive without evidence of PD were censored at the date of last disease assessment.
  The PFS results are based on data as of August 2012, while overall survival (OS) was updated in April 2014. Given the early termination and limited sample size, data management efforts to update PFS were not pursued.
Time Frame: Assessed every 3 months if patient is < 2 years from study entry, every 6 months if patient is 2-5 years from study entry, every 12 months if patient is 6-10 years from study entry, up to 10 years
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (VRD) | Arm B (VD)
Number analyzed (Participants) | 23 | 25
Months | NA [NA to NA] — Median PFS was not reached for Arm A (VRD). | 17.4 [7.1 to 35.4]
Statistical Analysis 1: Comparison: Arm A (VRD) vs Arm B (VD); Stratified log rank test was used to compare progression-free survival between the two arms; Test type: Superiority or Other; p = 0.092, Log Rank

2. Secondary Outcome: Response Rates (Complete Response [CR] or Very Good Partial Response [VGPR])
Description: CR:
  Patients with complete disappearance of an M-protein and no evidence of myeloma in the bone marrow are considered to have CR. To be considered CR, patients must meet all of the following criteria:
  * Negative immunofixation on the serum and urine at two consecutive times
  * Disappearance of any soft tissue plasmacytomas
  * ≤5% plasma cells in bone marrow
  * If serum and urine M protein are unmeasurable and the immunoglobulin free light chain (FLC) parameter is being used, patients must have a normal ratio of 0.26-1.65 at two consecutive times
  VGPR:
  * Serum and urine M-component detectable by immunofixation but not on electrophoresis OR
  * >=90% reduction in serum M-component plus urine M-component <100 mg per 24 hours (by SPEP and UPEP)
  * If the serum and urine M protein are unmeasurable and the immunoglobulin FLC parameter is being used, a >90% decrease in the difference between involved and uninvolved FLC levels is required in place of the M protein criteria
Time Frame: Assessed at the end of each cycle, every 3 months if patient is < 2 years from study entry, every 6 months if patient is 2-5 years from study entry, every 12 months if patient is 6-10 years from study entry, up to 10 years
Population: Patients with measurable disease at randomization were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of patients
Arm/Group | Arm A (VRD) | Arm B (VD)
Number analyzed (Participants) | 16 | 16
Proportion of patients | 0.625 [0.354 to 0.848] | 0.188 [0.041 to 0.457]
Statistical Analysis 1: Comparison: Arm A (VRD) vs Arm B (VD); Fisher's exact test was used to compare the response rates between the two arms; Test type: Superiority or Other; p = 0.029, Fisher Exact

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to death or date of last known alive. The OS results are based on data as of April 2014.
Time Frame: as for outcome 1
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (VRD) | Arm B (VD)
Number analyzed (Participants) | 23 | 25
Months | 64.0 [50.2 to 65.2] | NA [NA to NA] — Median overall survival was not reached in Arm B.
Statistical Analysis 1: Comparison: Arm A (VRD) vs Arm B (VD); Stratified log-rank test was used to compare overall survival between the two arms; Test type: Superiority or Other; p = 0.48, Log Rank

4. Secondary Outcome: Change in Quality of Life (QOL) From Baseline to 6 Months Post Consolidation as Assessed by the Functional Assessment of Cancer Therapy-Neurotoxicity Trial Outcome Index (FACT-Ntx TOI)
Description: The combined score on the FACT-Ntx TOI is of interest. The FACT-Ntx TOI has 25 items and the score ranges from 0 (worst possible quality of life) -100 (best possible quality of life). The primary QOL endpoint is defined as the change in the FACT-Ntx TOI score from registration to 6 months post consolidation treatment.
Time Frame: Baseline and 6 months post consolidation treatment
Population: Patients with both assessments complete at baseline and 6 months post consolidation treatment were included in this analysis.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Arm A (VRD) | Arm B (VD)
Number analyzed (Participants) | 12 | 8
units on a scale | -7.9 [-43.0 to 20.0] | -2.6 [-20 to 20]

ADVERSE EVENTS:
Time Frame: Assessed every 21 days while on treatment and for 30 days after the end of treatment
Groups:
- Arm A (VRd Regimen): Arm A (VRd Regimen) Patients were given consolidation therapy for 8 cycles (1 cycle = 21 days) with the combination bortezomib, dexamethasone and lenalidomide. Patients received each cycle: the standard dose of bortezomib (1.3 mg/m2) on days 1, 4, 8 and 11; fixed dose of lenalidomide at 15 mg orally on days 1-14; and 3 days of dexamethasone at 40 mg total dose per day given on days 1, 8 and 15. Aspirin 325 mg/day orally on days 1-21 of each cycle was required unless the patient was treated with alternate prophylaxis of either low molecular weight heparin or coumadin.
- Arm B (Vd Regimen): Arm B (Vd Regimen) Patients were given consolidation therapy for 8 cycles (1 cycle = 21 days) with the combination bortezomib plus dexamethasone. Patients received each cycle: the standard dose of bortezomib (1.3 mg/m2) on days 1, 4, 8 and 11 and 3 days of dexamethasone at 40 mg total dose per day given on days 1, 8 and 15.
Arm/Group | Arm A (VRd Regimen) | Arm B (Vd Regimen)
Serious Adverse Events (participants affected / at risk) | 15/23 | 16/25
Other Adverse Events (participants affected / at risk) | 8/23 | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (VRd Regimen) (N=23) | Arm B (Vd Regimen) (N=25)
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1
Leukocytes (Investigations) | 1 | 0
Lymphopenia (Investigations) | 3 | 1
Neutrophils (Investigations) | 0 | 2
Platelets (Investigations) | 2 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Fatigue (General disorders) | 3 | 4
Fever w/o neutropenia (General disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Infection w/ gr3-4 neut, lung (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, colon (Infections and infestations) | 0 | 2
Infection Gr0-2 neut, lung (Infections and infestations) | 1 | 1
ALT, SGPT (Investigations) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuropathy-motor (Nervous system disorders) | 2 | 0
Neuropathy-sensory (Nervous system disorders) | 6 | 6
Psychosis (Psychiatric disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 1 | 2
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Joint, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (VRd Regimen) (N=23) | Arm B (Vd Regimen) (N=25)
Hemoglobin (Blood and lymphatic system disorders) | 2 | 4
Leukocytes (Investigations) | 1 | 2
Lymphopenia (Investigations) | 1 | 3
Neutrophils (Investigations) | 0 | 2
Platelets (Investigations) | 1 | 4
Fatigue (General disorders) | 3 | 4
Insomnia (Psychiatric disorders) | 3 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1
Neuropathy-sensory (Nervous system disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less